CLINICAL TRIAL: NCT02743429
Title: Phase II Study of Monoclonal Antibody ch14.18/CHO Continuous Infusion in Patients With Primary Refractory or Relapsed Neuroblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medicine Greifswald (Other)
Collaborators: Children's Cancer Research Institute, Austria (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APN311-304; 2014-000588-42 (EudraCT Number)
Record Dates: First submitted 2016-03-18; First posted 2016-04-19 (Estimated); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Neuroblastoma
Keywords: ch14.18/CHO; neuroblastoma; long term infusion
MeSH Terms: conditions — Neuroblastoma | interventions — dinutuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Long term infusion of ch14.18/CHO (Experimental): 10 day continuous Infusion of ch14.18/CHO.
  Interventions: Drug: dinutuximab beta

INTERVENTIONS:
Drug: dinutuximab beta — Up to 5 cycles of continuous infusion of ch14.18/CHO is administered at a dose of 10 mg/m2/day over 10 days (total dose 100 mg/m2/cycle).
  Cycle duration: 35-days.

SUMMARY:
In this trial, monoclonal anti-Disialoganglioside GD2 (GD2) antibody ch14.18/CHO will be assessed for the treatment of patients with relapsed or refractory neuroblastoma. The antibody is used as a single agent applied in a new treatment schedule associated with less side effects.

DETAILED DESCRIPTION:
The Treatment with ch14.18 antibody has demonstrated efficacy in patients with neuroblastoma. However the treatment is associated with an on target side effect, i.e. neuropathic pain. This requires coadministration of intravenous morphine.

In this clinical Trial we will evaluate a less toxic treatment regimen consisting of continuous longterm Infusion (LTI) of ch14.18/CHO administered at a dose of 10 mg/m2/day over 10 days (total dose 100 mg/m2/cycle). Patients may receive up to five 35-day cycles in absence of signs of progression.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 12 months and ≤ 21 years of age at the time of study entry
2. Diagnosis of neuroblastoma according to the INSS criteria
3. Tumour burden controlled by conventional therapy (except patients with early minimal bone marrow relapse) fulfilling one of the following criteria:

   - Primary refractory patients with stage 4 disease
   * Relapse after primary stage 4 disease
   * Disseminated relapse after primary localized neuroblastoma.
4. Measurable and/or evaluable disease in any of the following sites (skeletal lesions, soft tissue lesions, lymph nodes and/or primary tumour site and/or bone marrow) as measured by mIBG scan, CT, MRI and/or immunocytology
5. Life expectancy of at least 12 weeks.
6. Performance status greater or equal to 70% (Lansky Score or Karnofsky)
7. Consent to the placement of a central venous line, if one has not already been placed
8. Off any standard or experimental treatment for at least two weeks prior to start of immunotherapy (Day 1 of cycle 1) and fully recovered from the short-term major toxic effects
9. No immediate requirements for palliative chemotherapy, radiotherapy or surgery
10. At least 2 weeks from any tumour surgery and fully recovered from any post-surgical complications
11. HIV sero-negative
12. Neither active nor chronic-replicative Hepatitis B infection
13. Females of childbearing potential must have a negative pregnancy test and must agree to use an effective birth control method during the whole study duration including the last FU visit.

    Female patients who are lactating must agree to stop breast-feeding.
14. Patient may have had prior CNS metastases, provided the following criteria are all met:

    * The patient's CNS disease has been previously treated.
    * The patient's CNS disease has been clinically stable for four weeks prior to starting this study (assessment must be made clinically and by CT or MRI).
    * The patient is off steroids for four weeks prior to starting trial treatment and will not require them during the course of the study.
15. Patients with seizure disorders may be enrolled if well controlled on anticonvulsants and if no seizures have occurred within a 6 week period prior to starting trial treatment
16. All patients and/or their parents or legal guardians must sign a written informed consent.
17. Laboratory testing:

    * Shortening fraction of ≥ 30% on Echocardiogram.
    * FEV1 and FVC > 60% of the predicted by pulmonary function tests. Children unable to do PFTs should have no dyspnoea at rest and a pulse oximetry > 94% in room air.
    * Adequate bone marrow function as defined by ANC >0.5 10^9/L, platelets ≥ 20 10^9/L and haemoglobin > 8.0 g/dL
    * Adequate liver function, as defined by an ALT or AST < 5 x normal and a total bilirubin < 1.0 mg/dL.
    * Adequate renal function, as defined by a serum creatinine <1.5 mg/dL or a creatinine clearance or radioisotope GFR of > 60 mL/minute/1.73 m².

Exclusion Criteria:

1. Progressive disease at the time of inclusion into the study.
2. ADA positivity due to previous treatment with an anti-GD2 antibody (e.g. ch14.18/SP2/0, ch14.18/CHO).
3. Previous treatment with ch14.18/CHO in this study.

e) Requirement, or likely requirement, for corticosteroids or other immunosuppressive drugs.

f) Concurrent treatment with any non-trial anticancer therapies. g) Patients with hypersensitivity against one component of the investigational product or against mouse proteins.

h) Female patients of childbearing potential if pregnant, nursing, or not using effective contraception during the treatment period, as the potential effects of ch14.18 on the fetus have not been determined.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03-27 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Anti-tumour activity of ch14.18/CHO continuous infusion | 2 years
  The response rate in patients with measurable/evaluable disease (skeletal lesions, soft tissue lesions, lymph nodes and/or primary tumour site and bone marrow) as measured by Metaiodobenzylguanidine scan (MIBG), Computed tomography (CT), Magnetic Resonance Imaging (MRI) and/or immunocytology at the end of the study.

SECONDARY OUTCOMES:
Progression-Free Survival | 5 years
Safety and tolerability | 2 years
  * Pain intensity and the need for appropriate medication for pain relief
  * Adverse events, vital signs and changes in clinical laboratory assessments
Immunogenicity | 2 years
  Immunogenicity: Anti-Drug Antibody (ADA)
Immunophenotyping | 2 years
  Unit: cells/µl
Antibody dependent cellular cytotoxicity (ADCC) | 2 years
  Unit: %
Complement dependent cytotoxicity (CDC) | 2 years
  Unit: %
Whole Blood Test (WBT) | 2 years
  Unit: %
Cytokines | 2 years
  Unit: µg/ml
Clearance (CL) | 2 years
  Unit: l/d*m²
Volume distribution at steady state (Vdss) | 2 years
  Unit: l/m²
mean residence time (MRT) | 2 years
  Unit: days
half-life time (t1/2) | 2 years
  Unit: days
Area Under the Curve (AUC) | 2 years
  Unit: µg*d/ml
Maximum Plasma Concentration (Cmax) and Minimum Plasma Concentration (Cmin) | 2 years
  Unit: µg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Holger Lode, Professor, Study Director — University Medicine Greifswald
Locations (2):
- St. Anna Kinderkrebsforschung e.V. CHILDREN'S CANCER RESEARCH INSTITUTE, Vienna, Austria
- University Medicine Greifswald, Greifswald, Germany

REFERENCES:
- [Derived] Lode HN, Ehlert K, Huber S, Troschke-Meurer S, Siebert N, Zumpe M, Loibner H, Ladenstein R. Long-term, continuous infusion of single-agent dinutuximab beta for relapsed/refractory neuroblastoma: an open-label, single-arm, Phase 2 study. Br J Cancer. 2023 Nov;129(11):1780-1786. doi: 10.1038/s41416-023-02457-x. Epub 2023 Oct 10. PMID 37813959